CLINICAL TRIAL: NCT04180397
Title: Goal Directed Fluid Removal With Furosemide in Intensive Care Patients With Fluid Overload - A Randomised, Blinded, Placebo-controlled Trial (GODIF).
Brief Title: Controlled Fluid Removal in Critical Ill Patients With Fluid Overload in the Intensive Care Unit.
Acronym: GODIF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Morten H. Bestle (Other)
Collaborators: University of Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Centre for Research in Intensive Care (CRIC) (Other)
Responsible Party: Sponsor-Investigator, Morten H. Bestle, Senior staff specialist and Professor, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GODIF
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Fluid Overload
Keywords: Fluid overload; Fluid removal; Deresusciation; Diuretics; Fluid accumulation
MeSH Terms: conditions — Edema | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide (Active Comparator): Bolus of 5-40 mg (0.5 - 4 ml) of furosemide iv at physicians discretion followed by infusion of furosemide. Infusion rate: 0-40 mg/hour. Starting rate: 20 mg/hour. The infusion is adjusted according effect. Target is a negative fluid balance of 1 ml/kg/hour. The fluid balance is calculated 3 times a dag at 6:00 am, 2:00 pm and 10:00 pm. Goal directed fluid removal is stopped when the fluid balance is assessed neutral.
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): Isotonic saline dosed the same way and by the same algorithm as for furosemide. Start bolus of 0.5-4 ml at physicians discretion. Infusion rate: 0 - 4 ml/hour. Infusion is started at 2 ml/hour and adjusted according to effect. Target is a negative fluid balance of 1 ml/kg/hour. The fluid balance is calculated 3 times a dag at 6:00 am, 2:00 pm and 10:00 pm. Goal directed fluid removal is stopped when the fluid balance is assessed neutral.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Furosemide — Furosemide 10 mg/ml for injection/infusion
  Other Names: Furix
  Arms: Furosemide
Drug: Isotonic saline — Isotonic saline used as placebo (injection/infusion)
  Arms: Placebo

SUMMARY:
This study evaluates the benefits and harms of goal directed fluid removal with furosemide versus placebo in critical ill adult patients with fluid overload in the intensive care unit. Half of the patients will receive furosemide and the other half placebo. The treatment will continue until the excess fluid is excreted.

DETAILED DESCRIPTION:
Fluid overload is a common and serious complication in patients admitted to the intensive care unit (ICU). A core element of therapy in the ICU is resuscitation with crystalloid solutions. In many cases fluid accumulate, and patients become fluid overloaded. Several observational studies indicate a detrimental effect of fluid overload in different clinical settings, including patients with acute kidney injury. It is unknown whether this association is causal or if the increased tendency to accumulate fluid is a marker of disease severity and thereby a higher risk of death. The investigators want to investigate this in critical ill patients with fluid overload of 5% or more by randomizing them to furosemide (diuretics) or placebo.

ELIGIBILITY:
Inclusion Criteria: ALL below must be met.

* Acute admission to the intensive care unit.
* Age ≥ 18 years of age
* Fluid overload ≥ 5% of ideal body weight. If possible, all fluids administered before admission to the intensive care unit are to be included in the calculation of cumulative fluid balance.
* Clinical stable (minimum criteria: MAP > 50 mmHg and maximum infusion of 20 microgram/kg/minute of noradrenaline and lactate < 4.0 mmol/L)

Exclusion Criteria:

* Known allergy to furosemide or sulphonamides.
* Known pre-hospitalization advanced chronic kidney disease (eGFR < 30 mL/minute/1.73 m^2 or chronic RRT).
* Ongoing renal replacement therapy.
* Anuria > 6 hours.
* Rhabdomyolysis with indication for forced diuresis
* Ongoing life-threatening bleeding as these patients need specific fluid/blood product strategies.
* Acute burn injury of more than 10% of the body surface area as these patients need a specific fluid strategy.
* Severe dysnatremia (p-Na < 120 or > 155 mmol/L) as these patients need a specific fluid strategy.
* Severe hepatic failure as per the clinical team.
* Patients undergoing forced treatment.
* Fertile women (women < 50 years) with positive urine human chorionic gonadotropin (hCG) or plasma-hCG.
* Consent not obtainable as per the model approved for the specific trial site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital | 90 days after randomization
  Days alive and out of hospital

SECONDARY OUTCOMES:
All cause mortality | 90 days after randomization
  All cause mortality
Mortality and life support | 90 days after randomization
  Days alive without life support without life support (vasopressor/inotropic support, invasive mechanical ventilation or renal replacement therapy)
Mortality 1 year | one year after randomization
  All cause mortality
Serious adverse events and reactions | 90 days
  Number of participants with one or more serious adverse events and serious adverse reactions
Health related quality of life | 1 year after randomization
  Measured using the European quality of Life 5D-5L questionnaire (5D-5L is the full name of the questionnaire). Index value of 1 represents full health and dead = 0. These value sets reflect the preferences of the general population. The European quality of life visual analogue scale is a self-reported assessment of the participant's health status. Scores on 100 = the best health you can imagine and 0 = the worst health you can imagine.
Cognitive function | 1 year after randomization
  Cognitive function assessed by the Montreal Cognitive Assessment score. Using the mini test for telephone interview. The test and scoring system will soon be published from Montreal Cognitive Assessment.
Health related quality of life | 1 year after randomization
  Subjective assessment (unacceptable, neutral, acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bestle, MD, Study Chair — Department of Anaesthesiology and Intensive Care medicine Nordsjællands hospital
Locations (24):
- Department of Intensive Care, Liverpool Hospital, Sydney, Australia
- Denmark (16):
  - Department of Intensive Care, Sygehus Sønderjylland Aabenraa, Aabenraa
  - Departmen of Intensive Care, Aalborg
  - Department of Intensive Care, Aarhus University Hospital, Aarhus
  - Department of Intensive Care, Rigshospitalet, Copenhagen
  - Departement of Intensive Care, Gentofte Hospital, Gentofte Municipality
  - Department of Intensive Care, Herlev Hospital, Herlev
  - Department of Intensive Care, Regionshospital Gødstrup, Herning
  - Department of Intensive Care, Nordsjællands hospital, Hillerød
  - Department of Intensive Care, Regionshospital Nordjylland Hjørring, Hjørring
  - Department of Intensive Care, Kolding
  - Department of Intensive Care, Zealand University hospital, Køge
  - Department of Intensive Care, Odense
  - Department of Intensive Care, Regionshospitalet Randers, Randers
  - Department of Intensive Care, University Hospital Zealand, Roskilde, Roskilde
  - Department of Intensive Care, Vejle
  - Regionshospitalet Viborg, Viborg
- Finland (2):
  - Department of Intensive Care, Tampere University Hospital, Tampere
  - Department of Intensive Care, Turku
- Department of Intensive Care, Landspitali National University Hospital of Iceland, Reykjavik, Iceland
- Department of Critical Care, University Medical Center Groningen, Groningen, Netherlands
- Norway (2):
  - Department of Intensive Care, Ålesund Sjukehus, Ålesund
  - Department of Intensive Care, Stavanger University Hospital, Stavanger
- Department of Intensive Care, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
will be made available on reasonable request after the primary results are published
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Wichmann S, Lange T, Perner A, Gluud C, Itenov TS, Berthelsen RE, Nebrich L, Wiis J, Brochner AC, Nielsen LG, Behzadi MT, Damgaard K, Andreasen AS, Strand K, Jarvisalo M, Strom T, Eschen CT, Vang ML, Hildebrandt T, Andersen FH, Sigurdsson MI, Thomar KM, Thygesen SK, Troelsen TT, Uusalo P, Jalkanen V, Illum D, Solling C, Keus F, Pfortmueller CA, Wahlin RR, Ostermann M, Aneman A, Bestle MH. Furosemide versus placebo for fluid overload in intensive care patients-The randomised GODIF trial second version: Statistical analysis plan. Acta Anaesthesiol Scand. 2024 Jan;68(1):130-136. doi: 10.1111/aas.14320. Epub 2023 Sep 11. PMID 37691474
- [Derived] Wichmann S, Itenov TS, Berthelsen RE, Lange T, Perner A, Gluud C, Lawson-Smith P, Nebrich L, Wiis J, Brochner AC, Hildebrandt T, Behzadi MT, Strand K, Andersen FH, Strom T, Jarvisalo M, Damgaard KAJ, Vang ML, Wahlin RR, Sigurdsson MI, Thormar KM, Ostermann M, Keus F, Bestle MH. Goal directed fluid removal with furosemide versus placebo in intensive care patients with fluid overload: A trial protocol for a randomised, blinded trial (GODIF trial). Acta Anaesthesiol Scand. 2022 Oct;66(9):1138-1145. doi: 10.1111/aas.14121. Epub 2022 Aug 9. PMID 35898170